CLINICAL TRIAL: NCT05197101
Title: To Evaluate the Efficacy and Safety of Balloon Catheter Combined With Oxytocin Induction in Nulliparous Women With Estimated Fetal Weight ≥3500g at 39-40 Weeks of Gestation: a Randomized, Controlled, Observational Study
Brief Title: To Evaluate the Efficacy and Safety of Balloon Catheter Combined With Oxytocin Induction in Nulliparous Women With Estimated Fetal Weight ≥3500g at 39-40 Weeks of Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PIIM
Record Dates: First submitted 2022-01-17; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Macrosomia, Fetal
Keywords: balloon catheter; oxytocin
MeSH Terms: conditions — Fetal Macrosomia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nulliparous women with estimated fetal weight ≥3500g at 39-40 weeks of gestation (Experimental)
  Interventions: Procedure: balloon catheter combined with oxytocin induction

INTERVENTIONS:
Procedure: balloon catheter combined with oxytocin induction — Balloon catheter for 12 hours and oxytocin for up to 3days.If failed , they will be treated ceacrean.

SUMMARY:
This study is a randomized, controlled, observational study. 150 nulliparous women with estimated fetal weight ≥3500g at 39-40 weeks of gestation will be enrolled as subjects in the two groups is 1:1. In the experimental group, vaginal examination will be performed at 39 to 40 weeks to assess cervical conditions. If the bishop score <6, the balloon catheter combined with oxytocin induction will be planned at 40 weeks ±3 days. In the control group, one week to 41 weeks ±3 days will be expected. Vaginal examination will be performed again to evaluate cervical conditions. If the bishop score <6 points, and balloon catheter combined with oxytocin induction will be performed. After 96h, their final delivery mode will be recorded. In the following 42 days postpartum, their complications and the neonatal outcome will be followed up.

ELIGIBILITY:
Inclusion Criteria: singleton head position pregnancy, negative Down's screening and /or NIPT screening, no malformation was found, with slight/without pregnancy complications -

Exclusion Criteria:twin or multiple pregnancy, scar uterus, with contraindications to vaginal delivery, estimated fetal weight >4500g

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-01-17 (Estimated); Primary Completion 2023-01-17 (Estimated); Study Completion 2023-03-17 (Estimated)

PRIMARY OUTCOMES:
vaginal birth rate | 24 hours
  After spontaneous labor for up tp 24 hous, the mode of delivery will be konwn and recorded.

IPD SHARING:
Plan to Share IPD: Undecided